CLINICAL TRIAL: NCT06700356
Title: Seizure Detection With a Deep Brain Stimulation System
Brief Title: Thalamus Seizure Detection With a Deep Brain Stimulator System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Nicholas Gregg, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-012058
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Epilepsy; Seizure
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Thalamus seizure detection with a DBS system (Experimental): Thalamus seizure detection by a DBS system, validated with concurrent in-hospital gold standard video EEG monitoring.
  Interventions: Device: Phase 1-Validation of thalamus seizure detection with concurrent video EEG monitoring; Device: Phase 2-DBS Stimulation with Medtronic Percept DBS device-Out Patient

INTERVENTIONS:
Device: Phase 1-Validation of thalamus seizure detection with concurrent video EEG monitoring — Epilepsy monitoring unit evaluation will follow standard of care practices for seizure characterization, and antiseizure medications may be reduced to facilitate the recording of seizures. Patient clinical management, and video-EEG interpretation will be completed by the clinical epilepsy monitoring unit team which consists of physicians, nurse practitioners, registered nurses, and in-house 24-hour 7-days-per-week EEG technicians. Continuous full-bandwidth thalamus recordings (250 Hz) will be acquired by the research study team using a standard clinician programmer and telemetry module. Hospital monitoring will last up to 4 days.
Device: Phase 2-DBS Stimulation with Medtronic Percept DBS device-Out Patient — Patients will then transition to the ambulatory phase. In the outpatient setting, patients will have constrained ambulatory thalamus recordings using recording parameters determined by Phase 1. DBS treatment stimulation will be programmed in the clinical epilepsy neuromodulation lab using typical high frequency (>50 Hz) stimulation. High frequency stimulation is the conventional approach to DBS for epilepsy, as was used in the pivotal study leading to premarket approval (SANTE study)2 of anterior nucleus of the thalamus (ANT) DBS for focal epilepsy, which is typical for epilepsy DBS practice3, and several studies of DBS for generalized epilepsy4-6, in a sensing friendly electrode configuration. Patients will keep a detailed seizure diary. Ambulatory thalamus recordings by the DBS system and patient reported seizure diaries will be collected during routine clinical DBS programming visits (q3-9 months).

SUMMARY:
The purpose of this study is to determine the feasibility of chronic ambulatory thalamus seizure detection. The sensitivity, specificity, and false alarm rate of thalamus seizure detection will be calculated using recordings from a deep brain stimulation system, assessed relative to concurrent gold-standard video-EEG monitoring collected in the in-patient setting (epilepsy monitoring unit), in 5 patients with drug resistant epilepsy.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the inclusion criteria to participate in this study:

* 18 years of age and older.
* Implanted with a clinical DBS system for epilepsy with brain recording capabilities (Medtronic Percept™ DBS).
* Subject or legally authorized representative is able to understand study procedures and to comply with them for the entire length of the study.

Exclusion Criteria:

All candidates meeting any of the exclusion criteria at baseline will be excluded from study participation:

* Health status or any clinical conditions (e.g., life expectancy, co-existing disease) that, in the opinion of the site investigator, would pose undue risk to undergo epilepsy monitoring unit evaluation for the purpose of seizure characterization.
* Women will verify not pregnant, and if applicable, have urine pregnancy test.
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Thalamic seizure detection in the epilepsy monitoring unit | 2 years
  The sensitivity, specificity, and false alarm rate of thalamus seizure detection will be calculated using recordings from a deep brain stimulation system, assessed relative to concurrent gold-standard video-EEG monitoring collected in the epilepsy monitoring unit, in patients with drug resistant epilepsy.

SECONDARY OUTCOMES:
Ambulatory thalamus seizure detection with constrained DBS recordings | 2 years
  The sensitivity, specificity, and false alarm rate of chronic ambualtory thalamus seizure detection will be calculated using constrained local field potential power-in-band recordings from a deep brain stimulation system, assessed relative to patient reported seizure diary.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Gregg, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No